CLINICAL TRIAL: NCT03573141
Title: The Relationship of Manual Physical Therapy to Habitual Physical Activity and Sleep Behavior for Patients With Knee Osteoarthritis
Brief Title: Influence of Manual Physical Therapy on Habitual Activity in Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nathan Parsons, Principal Investigator, Fellow-in-Training, Army-Baylor Doctoral Fellowship in Orthopedic Manual Physical Therapy, Brooke Army Medical Center
Other Study IDs: C.2017.167
Record Dates: First submitted 2018-05-15; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee OA patients receiving Physical Therapy: Only 1 group was included in this study. Subject's physical activity and sleep quality were assessed at baseline, prior to treatment. Follow up data was collected immediately after a course of physical therapy then again 8 weeks later.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Subjects received a comprehensive physical therapy evaluation after baseline data collection and received a normal course pf physical therapy treatment based on impairments identified.

SUMMARY:
The investigators assessed overall physical activity and sleep quality in subjects with knee osteoarthritis(OA) at baseline, and at four and 12 weeks following initiation of physical therapy. Subjects received a course of manual physical therapy with interventions targeted to relevant impairments in the lower quarter. No progressive activity intervention or guidance on sleep hygiene was included. The purpose of this study was to assess a relationship between manual physical therapy and habitual physical activity and sleep behavior in individuals with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Knee pain and crepitus with active motion and morning stiffness < 30 minutes and age > 38 years old.
2. Knee pain and crepitus with active motion and morning stiffness < 30 minutes and bony enlargement.
3. Knee pain and no crepitus and bony enlargement.

Participants will have to meet all of the following additional inclusion criteria:

1. Age > 38 years old.
2. Tricare beneficiary
3. Ability to read and speak English well enough to provide informed consent and follow study instructions
4. Knee OA is the participant's most physically limiting condition as determined by patient's self report.
5. Able to ambulate 20 meters (65.6 feet) feet without an assistive device.
6. Radiographic findings of knee OA

Exclusion Criteria:

* 1.) Presence of any medical "Red Flags" affecting the knee:

  1. Tumor, neoplasm etc. affecting the knee
  2. Current or past history of rheumatoid arthritis or similar rheumatic condition
  3. Current or past history of gout or pseudogout affecting the knee
  4. Active Infection in the knee within the past 12 months

     2.) Inability to participate in the therapy plan prescribed by the treating therapist 3.) Any prior Physical Therapy for the knee in the past 12 months 4.) Injection to the knee joint within the previous 30 days 5.) Surgical procedure on either lower extremity within the past 6 months 6.) Any prior lower extremity joint replacement surgery 7.) A physical impairment unrelated to the knee that prevents the subject from safely participating in any aspect of the study 8.) History of cardiac, respiratory, or musculoskeletal disorders (e.g. amputation) that restrict lower extremity function. 9.) Any physical, psychological, or emotional condition that is more symptom producing, or activity limiting than their knee OA.

     10.) Any condition that disrupts sleep more than knee OA, such as a sleep disorder or Obstructive Sleep Apnea 11.) Inability to speak/read English adequately to understand and provide informed consent 12.) Pregnant or intending to become pregnant in the next year 13.) Military service members in a WTU (Warriors in Transition Unit) or service equivalent or pending a medical evaluation board/discharge process. For non-military personnel, anyone that is pending or undergoing any litigation. 14.) WOMAC Score < 30 15.) Unable to provide informed consent to participate in the study

Age Groups: Child, Adult, Older Adult
Study Population: Military Retirees and dependents receiving care for primary diagnosis of knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Total Steps Per Day from baseline to 4 weeks and 12 weeks | 1 week of monitoring at baseline, 4 weeks and 12 weeks
  Steps per day were measured with an ActiGraph accelerometer (model wGT9X Link), ActiGraph Corp., Pensacola FL). The ActiGraph accelerometer measures triaxial acceleration and provides information about the intensity and duration of the physical activity associated with movement.
Change in Total Sedentary Time from baseline to 4 weeks and 12 weeks | 1 week of monitoring at baseline, 4 weeks and 12 weeks
  Total Sedentary Time was measured with an ActiGraph accelerometer (model wGT9X Link), ActiGraph Corp., Pensacola FL). The ActiGraph accelerometer measures triaxial acceleration and provides information about the intensity and duration of the physical activity associated with movement. Total time spent in sedentary was calculated based on established on established cut points, reported in minutes per day and converted to a percentage of daily activity. Higher percentage indicated more time spent in sedentary behavior.
Change in Sleep Efficiency from baseline to 4 weeks and 12 weeks | 1 week of monitoring at baseline, 4 weeks and 12 weeks
  Sleep efficiency is defined as the total sleep time relative to the time in bed. Higher scores indicated better sleep efficiency, with scores above 85 considered to be in the normal range. Sleep monitoring was performed using the Micro Motionlogger Sleep Watch (Ambulatory Monitoring Inc., Ardsley, NY) on the non-dominant wrist.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) from baseline to 4 weeks and 12 weeks | Collected at baseline, 4 weeks and 12 weeks
  The primary patient-reported outcome was the Western Ontario and McMaster's University Arthritis Index(WOMAC). It is a widely used, proprietary standardized questionnaire used by health professionals to evaluate the condition of patients with OA of the knee and hip, including pain, stiffness, and physical functioning. This scale runs from 0 to 240 points with lower scores indicating improved symptoms and function.

SECONDARY OUTCOMES:
Change in 400-meter walk time from baseline to 4 weeks and 12 weeks | Collected at baseline, 4 weeks and 12 weeks
  The 400-meter walk test was administered to quantify walking endurance. The test was conducted a 100-meter-long course with four lengths being completed. Timing using a digital stopwatch began from the initial movement from standing at the start until the subject completed the fourth length of the course. Total time (sec) was recorded, with longer time indicating worse physical function
Change in 20-meter walk time from baseline to 4 weeks and 12 weeks | Collected at baseline, 4 weeks and 12 weeks
  The 20-meter walk test was performed in a hallway located in the PT Clinic which was free from any potential barriers to ambulation. The 20-meter walk course was clearly marked with bright cones at each end. Participants were instructed to wear their regular footwear and to use any assistive devices they normally use for ambulation. Total time (sec) was recorded and converted to meters per second, with a lower value indicating worse physical function.
Change in Timed Up and Go (TUG) time from baseline to 4 weeks and 12 weeks | Collected at baseline, 4 weeks and 12 weeks
  The TUG is a simple test of mobility designed to assess dynamic balance. Participants were expected to wear their regular footwear and use any assistive devices they normally use for ambulation. Total time (sec) was recorded with a lower value indicating worse physical function.
Change in Five Times Sit to Stand(5TSTS)time from from baseline to 4 weeks and 12 weeks | Collected at baseline, 4 weeks and 12 weeks
  The 5TSTS was used to determine lower extremity functional strength. Participants were instructed to stand from a chair and return to sitting five times as quickly as possible with arms folded across the chest. Total time in seconds was measured with a digital stopwatch and started with initial movement to stand on the first repetition and ended after completely standing upright on the 5th repetition, with longer time indicating worse physical function
Change in acceleration while stepping off a curb from baseline to 4 weeks and 12 weeks | Collected at baseline, 4 weeks and 12 weeks
  Vertical acceleration forces were measured with Shimmer3 monitors (Shimmer Sensing, Dublin, Ireland) at the waist and lower leg in order to assess instrumented evaluation of stepping off a raised platform while walking. This task is ubiquitous in daily activity throughout the lifespan. There is no greater risk with this test than stepping off a typical curb. Participants completed the task under close supervision by research staff by stepping down from a 20 cm raised platform in the PT clinic to simulate a curb. 5 trials were completed with both lower extremities at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Jennifer Moreno Clinic, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No